CLINICAL TRIAL: NCT03534960
Title: High Flow Nasal Oxygen Therapy in Pediatric Hypercapnic Respiratory Failure During Perioperative Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Bin He, Associate Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-17-007
Record Dates: First submitted 2017-07-23; First posted 2018-05-23 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High Flow Nasal Oxygen Therapy (Other): Patients are randomized to the high flow nasal oxygen therapy group
  Interventions: Device: High Flow Nasal Oxygen Therapy
- Nasal CPAP (Other): Patients are randomized to the nasal continuous positive airway pressure treatment group
  Interventions: Device: Nasal CPAP

INTERVENTIONS:
Device: High Flow Nasal Oxygen Therapy — Nasal cannula flows of 3 to 8 lpm via systems approved to provide increased humidification and warmth to inspired gas
  Arms: High Flow Nasal Oxygen Therapy
Device: Nasal CPAP — Standard nasal CPAP via "bubble" or ventilator support at levels of 4-8 cm H2O
  Arms: Nasal CPAP

SUMMARY:
Humidified high flow nasal oxygen therapy decreases dilution of the inhaled oxygen and, by matching patient's peak flow, allows accurate delivery of the set FiO2 throughout the whole inspiratory phase.The purpose of this study is to determine the impact of hign-flow nasal therapy on pediatric hypercapnic respiratory failure by comparing with nasal continuous positive airway pressure.

DETAILED DESCRIPTION:
Humidified high flow nasal oxygen therapy decreases dilution of the inhaled oxygen and, by matching patient's peak flow, allows accurate delivery of the set FiO2 throughout the whole inspiratory phase.The purpose of this study is to determine the impact of hign-flow nasal therapy on pediatric hypercapnic respiratory failure by comparing with nasal continuous positive airway pressure

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from 1 to 18 years
2. Hypercapnic respiratory failure:

   PaO2<60mmHg and PaCO2 >50 mmHg
3. Candidate for non-invasive respiratory support as a result of:

   1. an intention to manage the patient with non-invasive (no endotracheal tube) respiratory support
   2. an intention to extubate the patient being managed with intubated respiratory support to non-invasive support

Exclusion Criteria:

1. Participation in a concurrent study that prohibits the use of HHFNC
2. Active air leak syndrome
3. Patients with abnormalities of the upper and lower airways; such as Pierre- Robin, Treacher-Collins, Goldenhar, choanal atresia or stenosis,
4. Patients with significant abdominal or respiratory malformations including tracheo-esophageal fistula, intestinal atresia, omphalocele, gastroschisis, and congenital diaphragmatic hernia
5. PaCO2<50mmHg

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-13 (Actual); Primary Completion 2018-11-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the number of patients in each group who require endotracheal intubation w | 24 hours

SECONDARY OUTCOMES:
mechanical ventilation-free to day 28 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided